CLINICAL TRIAL: NCT01650077
Title: Early Assessment of Therapeutic Response of Patients With Soft Tissue Sarcoma According to CHOI Criteria: Retrospective Study of Feasibility
Brief Title: Therapeutic Response of Patients With Soft Tissue Sarcoma According to CHOI Criteria
Acronym: ProAcTyon
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: ProAcTyon - 1203
Record Dates: First submitted 2012-07-19; First posted 2012-07-26 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma; Yondelis; Intolerance to doxorubicin/ifosfamide; CHOI criteria
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Non-interventional study consisting of a population of patients who had received for soft tissue sarcoma by at least 2 courses of Yondelis® at a dose of 1.5 mg / m² / 3 weeks after failure or intolerance to doxorubicin / ifosfamide from 2007 to 2011.

DETAILED DESCRIPTION:
Patient selection is based on a database of retrospectively within the GSF / GETO.

The tumor assessment must be made by scanner at baseline and post-C2 or C3 and should be available and sent to sponsor.

The comparative reading of the imaging is centralized and made without the knowledge of the local assessment:

* sum of the large diameter for 2 imagery (baseline and 1st evaluation
* tumor density on areas of interest for the 2 imaging (baseline and 1st evaluation
* Rank patients according to two methods (Choi and RECIST): complete response, partial response, stability, progress and non-assessable.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* locally advanced or metastatic soft tissue sarcoma
* treated with Yondelis after failure or intolerance to doxorubicin/ifosfamide
* treated between 2007 and 2011
* have had at least 2 cycles of Yondelis
* assessment of tumor by CT scan (baseline and after 2 or 3 cycles of Yondelis)

Exclusion Criteria:

* Gastro Intestinal Stromal Tumor GIST
* primitive bone sarcoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with soft tissue sarcoma treated with at least 2 cycles of Yondelis after failure or intolerance to doxorubicin/ifosfamide
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2012-09-21 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-10-28 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of tumor response according to CHOI criteria | after 6 weeks of treatment
  percentage of cases with a feasible evaluation according to CHOI

SECONDARY OUTCOMES:
To classify patients into two categories (progression or no progression) according to RECIST and to CHOI | after 6 weeks of treatment
  percentage of cases with a feasible evaluation according to RECIST
To determine percentage of false progression | after 6 weeks of treatment
  define as patient progressing according to RECIST and not progressing according to CHOI number of patient in each categories, according to each method of measurement
To determine predictive values of progression free survival and overall survival | after 6 weeks of treatment
  progression free survival = median time between date of inclusion and date of clinical or radiological progression overall survival = median time between date of inclusion and date of death
To characterize the profile of patients in false progression | after 6 weeks of treatment
  patient in progression according to RECIST but not progressing according to CHOI

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PENEL, MD, Study Director — Oscar Lambret Center
Locations (6):
- France (6):
  - Bergonie Institute, Bordeaux
  - Oscar Lambret Center, Lille
  - Antoine Lacassagne Center, Nice
  - Curie Institute, Paris
  - Henri Becquerel Center, Rouen
  - Cancer Institute of the West, Saint-Herblain